CLINICAL TRIAL: NCT02238509
Title: A Randomised, Multicentre, Open-label Phase II Trial Investigating Activity of Chemotherapy and Lapatinib and Trastuzumab in Patients With HER2-positive Metastatic Breast Cancer (MBC) Refractory to Anti HER2 Therapies
Brief Title: Safety and QoL of Trastuzumab With Lapatinib or Chemiotherapy in MBC and HER2+ Patients Refractory to Anti HER2 Therapies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorzio Oncotech (Other)
Collaborators: Clinical Research Technology S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIM12-TYPHER; 2013-005044-29 (EudraCT Number)
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; HER2 Positive; HER2+; MBC; Metastatic; Metastatic breast cancer; Chemotherapy; Lapatinib; Trastuzumab; anti HER2 therapies
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Lapatinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lapatinib and trastuzumab (Experimental): ARM A: Lapatinib and trastuzumab (experimental arm). Patients with hormone receptor (HR) positive breast cancer will also receive endocrine therapy at the physician's discretion (preferred choice with fulvestrant).
  Interventions: Drug: Lapatinib; Drug: Trastuzumab
- trastuzumab plus chemotherapy (Experimental): ARM B: Trastuzumab plus chemotherapy (control arm). Any type of chemotherapy in combination with trastuzumab will be allowed at the physician's discretion.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Lapatinib — ARM A: oral lapatinib 1,000 mg daily in combination with intravenous trastuzumab 6mg/kg q3wks (after the initial 8 mg/kg loading dose).
  Other Names: Tyverb
  Arms: lapatinib and trastuzumab
Drug: Trastuzumab — ARM A: oral lapatinib 1,000 mg daily in combination with intravenous trastuzumab 6mg/kg q3wks (after the initial 8 mg/kg loading dose).
  Other Names: Herceptin

SUMMARY:
Recent clinical studies have shown that the combination of lapatinib and trastuzumab has superior antitumor activity compared to either single drug in both neoadjuvant and metastatic setting and is well tolerated. According to this evidence, the combination of lapatinib and trastuzumab today offers a valid chemotherapy-free option, primarily for patients with pre-treated HER2-positive MBC

DETAILED DESCRIPTION:
The present study is designed to determine the efficacy and safety profile of the combination of lapatinib and trastuzumab (plus endocrinetherapy in ER-positive breast cancer) versus trastuzumab and chemotherapy in heavily pretreated patient population with HER2-positive MBC and to investigate the predictive role of cfDNA for detection of HER2 gene amplification on patients' outcome. The presence of circulating free DNA (cfDNA) for detection of HER2 gene amplification was associated with worse prognosis and seems to allow early response evaluation. However, many aspects of the role of cfDNA detection in patients undergoing molecular target agents such as trastuzumab or lapatinib are not well described. With the availability of improved and standardized techniques for cfDNA detection, it should now be possible to examine several of these important questions within a prospective multicenter study and a striking potential of cfDNA for detection of HER2 gene amplification might enable a more individual and optimized antimetastatic therapy inpatients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed and documented adenocarcinoma of the breast with metastatic disease
* The original tumour specimen must be HER2 IHC 3+ positive or, in case of IHC 2+
* Age ≥18
* Life expectancy of >12 weeks
* ECOG PS 0-1
* Measurable disease as defined by RECIST1.1 criteria
* All patients must have received prior anthracycline-and taxane-based regimens as well as trastuzumab based regimens in either the adjuvant or the metastatic setting. Patients must have been already treated with at least one line of the anti HER2 inhibitor therapy lapatinib for their metastatic breast cancer. A maximum of three previous lines of anti-HER-2 therapies in the metastatic setting are allowed.
* Adequate haematological function as defined by: ANC 1.5 x 109/L, platelet count 100 x 109/L, haemoglobin 10 g/dL.
* Adequate renal function, as defined by: creatinine 1.5 x UNL
* Adequate hepatobiliary function, as defined by the following baseline liver function tests: total serum bilirubin 1.5 upper normal limit (UNL); alanine amino transferase (ALT), aspartate amino transferase (AST) 2.5xUNL; alkaline phosphatase (AP) 2.5xUNL; if total alkaline phosphatase (AP) > 2.5xUNL, alkaline phosphatase liver fraction must be 2.5xUNL
* Adequate contraception for all fertile patients
* Negative pregnancy test.
* Postmenopausal women fulfilling any of the NCCN criteria may be included.
* Left ventricular ejection fraction (LVEF) ≥50% during a baseline period of 28 days, as determined by either echocardiography (ECHO) or multi gated acquisition (MUGA) scan.
* Signed, written informed consent

Exclusion Criteria:

* History of persistent Grade ≥ 2 hematologic toxicity resulting from previous systemic therapy
* Current peripheral neuropathy of NCI-CTCAE, Version 3.0, Grade ≥ 3 at randomization
* History of other malignancy within the last 5 years, except for carcinoma in situ of the cervix or basal cell carcinoma
* Bone-only disease, unless a measurable lesion is evident as determined by RECIST v1.1
* Bone scan, PET scan or plain films are not considered adequate imaging techniques to measure bone lesions. ve
* Blastic bone lesions are non-measurable.
* Uncontrolled hypertension (systolic >150 mm Hg and/or diastolic >100 mm Hg) or clinically significant (i.e. active) cardiovascular disease.
* Current dyspnoea at rest due to complications of advanced malignancy, or other diseases that require continuous oxygen therapy.
* Inadequate organ function, evidenced by the following laboratory results within 28 days prior to randomization.
* Current severe, uncontrolled systemic disease
* Major surgical procedure or significant traumatic injury within 28 days prior to study treatment start or anticipation of the need for major surgery during the course of study treatment
* History of receiving any investigational treatment within 28 days of randomization
* Current known infection with HIV, HBV, or HCV
* Receipt of IV antibiotics for infection within 14 days of randomization
* Known hypersensitivity to any of the study drugs
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol
* Lack of physical integrity of the upper gastrointestinal tract, clinically significant malabsorption syndrome, or inability to take oral medications
* Concurrent interventional or non-interventional studies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Rate | Clinical Benefit Rate is defined as confirmed complete response plus partial response at any time, plus stable disease up to 24 weeks
  To evaluate clinical benefit rate (CBR) for patients treated with lapatinib and trastuzumab and for patients treated with trastuzumab and chemotherapy. CBR is defined as: confirmed complete response (CR) plus partial response (PR) at any time, plus stable disease (SD) for 24 weeks

SECONDARY OUTCOMES:
Progression free survival | Patients enrolled will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever comes first, assessed up to 36 months
  Second-line progression-free survival, defined as the time from first dosing to the first documented disease progression or death from any cause, whichever occurs first.
Overall Survival | Patients enrolled will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever comes first, assessed up to 36 months
  OS is defined as the time from first dosing in second line to death from any cause.
Safety and tolerability | Patients enrolled will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever comes first, assessed up to 36 months
  Safety of second line treatment will be evaluated by the frequency of AEs and SAEs, cardiac events, clinically significant abnormal laboratory tests, vital signs, and ECOG PS. All patients who received at least one dose of study treatment will be included in the safety analysis.
Quality of life | Patients enrolled will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever comes first, assessed up to 36 months
  QoL and symptom control will be assessed using the FACT-B questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Grazia Arpino, MD, Principal Investigator — Dipartimento di Medicina Clinica e Chirurgia Oncologia Università degli Studi di Napoli "Federico II"
Locations (36):
- Italy (36):
  - A.O.U. Ospedali Riuniti Umberto I, Ancona
  - Centro di Riferimento Oncologico, Aviano
  - Policlinico S. Orsola Malpighi, Bologna
  - Ospedale Centrale di Bolzano, Bolzano
  - Presidio Ospedaliero 'Antonio Perrino, Brindisi
  - A.O.R.N.A.S. Garibaldi Nesima di Catania, Catania
  - Humanitas Centro Catanese di Oncologia, Catania
  - Azienda Ospedaliera S. Anna, Como
  - Ospedale 'F. Spaziani', Frosinone
  - I.R.C.C.S. A.O.U. San Martino, Genova
  - Ospedale Civile di Guastalla, Guastalla
  - Ospedale Vito Fazzi, Lecce
  - Ospedale di Lugo - AUSL della Romagna, Lugo
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Ospedale Niguarda Ca' Granda, Milan
  - A.O. San Gerardo, Monza
  - AORN "A. Cardarelli", Naples
  - Istituto Nazionale Tumori - IRCCS "Fondazione G.Pascale", Napoli
  - Policlinico SUN, Napoli
  - Università degli Studi di Napoli "Federico II", Napoli
  - A.R.N.A.S. Ospedale Civico e Benfratelli, Palermo
  - Ospedale S. Maria della Misericordia, Perugia
  - Azienda Ospedaliera Santa Maria degli Angeli, Pordenone
  - Ospedale di Ravenna, Ravenna
  - Arcispedale S. Maria Nuova Azienda Ospedaliera di Reggio Emilia, Reggio Emilia
  - Ospedale Infermi di Rimini, Rimini
  - Policlinico Universitario Campus Biomedico, Roma
  - Istituto Regina Elena per lo studio e la cura dei tumori, Roma
  - Ospedale G. Da Procida, Salerno
  - Ospedale Civile di Sassari SS Annunaziata, Sassari
  - Ospedale 'SS. Trinità', Sora
  - Azienda Ospedaliera S.Maria di Terni, Terni
  - A.O.U. San Giovanni Battista di Torino, Torino
  - A.O.U. Santa Maria della Misericordia di Udine, Udine
  - A.O. Ospedale di Circolo e Fondazione Macchi, Varese
  - Ospedale Sacro Cuore Don Calabria, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nahta R, Esteva FJ. Herceptin: mechanisms of action and resistance. Cancer Lett. 2006 Feb 8;232(2):123-38. doi: 10.1016/j.canlet.2005.01.041. PMID 16458110
- [Background] Nahta R, Yu D, Hung MC, Hortobagyi GN, Esteva FJ. Mechanisms of disease: understanding resistance to HER2-targeted therapy in human breast cancer. Nat Clin Pract Oncol. 2006 May;3(5):269-80. doi: 10.1038/ncponc0509. PMID 16683005
- [Background] Jagiello-Gruszfeld A, Tjulandin S, Dobrovolskaya N, Manikhas A, Pienkowski T, DeSilvio M, Ridderheim M, Abbey R. A single-arm phase II trial of first-line paclitaxel in combination with lapatinib in HER2-overexpressing metastatic breast cancer. Oncology. 2010;79(1-2):129-35. doi: 10.1159/000318043. Epub 2010 Nov 22. PMID 21088439
- [Background] Geyer CE, Forster J, Lindquist D, Chan S, Romieu CG, Pienkowski T, Jagiello-Gruszfeld A, Crown J, Chan A, Kaufman B, Skarlos D, Campone M, Davidson N, Berger M, Oliva C, Rubin SD, Stein S, Cameron D. Lapatinib plus capecitabine for HER2-positive advanced breast cancer. N Engl J Med. 2006 Dec 28;355(26):2733-43. doi: 10.1056/NEJMoa064320. PMID 17192538
- [Background] Clemens M, Eidtmann H, Nitz U, Niederle N, du Bois A, Grischke EM, Hinke A, von Minckwitz G. Trastuzumab single-drug therapy after failure of cytotoxic treatment for metastatic breast cancer. Onkologie. 2010;33(8-9):425-30. doi: 10.1159/000318144. Epub 2010 Jul 27. PMID 20838057
- [Background] von Minckwitz G, Schwedler K, Schmidt M, Barinoff J, Mundhenke C, Cufer T, Maartense E, de Jongh FE, Baumann KH, Bischoff J, Harbeck N, Luck HJ, Maass N, Zielinski C, Andersson M, Stein RC, Nekljudova V, Loibl S; GBG 26/BIG 03-05 study group and participating investigators. Trastuzumab beyond progression: overall survival analysis of the GBG 26/BIG 3-05 phase III study in HER2-positive breast cancer. Eur J Cancer. 2011 Oct;47(15):2273-81. doi: 10.1016/j.ejca.2011.06.021. Epub 2011 Jul 7. PMID 21741829
- [Background] Blackwell KL, Burstein HJ, Storniolo AM, Rugo H, Sledge G, Koehler M, Ellis C, Casey M, Vukelja S, Bischoff J, Baselga J, O'Shaughnessy J. Randomized study of Lapatinib alone or in combination with trastuzumab in women with ErbB2-positive, trastuzumab-refractory metastatic breast cancer. J Clin Oncol. 2010 Mar 1;28(7):1124-30. doi: 10.1200/JCO.2008.21.4437. Epub 2010 Feb 1. PMID 20124187
- [Background] Wu Y, Amonkar MM, Sherrill BH, O'Shaughnessy J, Ellis C, Baselga J, Blackwell KL, Burstein HJ. Impact of lapatinib plus trastuzumab versus single-agent lapatinib on quality of life of patients with trastuzumab-refractory HER2+ metastatic breast cancer. Ann Oncol. 2011 Dec;22(12):2582-2590. doi: 10.1093/annonc/mdr014. Epub 2011 Mar 15. PMID 21406472
- [Background] Johnston S, Pippen J Jr, Pivot X, Lichinitser M, Sadeghi S, Dieras V, Gomez HL, Romieu G, Manikhas A, Kennedy MJ, Press MF, Maltzman J, Florance A, O'Rourke L, Oliva C, Stein S, Pegram M. Lapatinib combined with letrozole versus letrozole and placebo as first-line therapy for postmenopausal hormone receptor-positive metastatic breast cancer. J Clin Oncol. 2009 Nov 20;27(33):5538-46. doi: 10.1200/JCO.2009.23.3734. Epub 2009 Sep 28. PMID 19786658
- [Background] Page K, Hava N, Ward B, Brown J, Guttery DS, Ruangpratheep C, Blighe K, Sharma A, Walker RA, Coombes RC, Shaw JA. Detection of HER2 amplification in circulating free DNA in patients with breast cancer. Br J Cancer. 2011 Apr 12;104(8):1342-8. doi: 10.1038/bjc.2011.89. Epub 2011 Mar 22. PMID 21427727
- [Background] Romond EH, Perez EA, Bryant J, Suman VJ, Geyer CE Jr, Davidson NE, Tan-Chiu E, Martino S, Paik S, Kaufman PA, Swain SM, Pisansky TM, Fehrenbacher L, Kutteh LA, Vogel VG, Visscher DW, Yothers G, Jenkins RB, Brown AM, Dakhil SR, Mamounas EP, Lingle WL, Klein PM, Ingle JN, Wolmark N. Trastuzumab plus adjuvant chemotherapy for operable HER2-positive breast cancer. N Engl J Med. 2005 Oct 20;353(16):1673-84. doi: 10.1056/NEJMoa052122. PMID 16236738
- [Background] Wang YC, Morrison G, Gillihan R, Guo J, Ward RM, Fu X, Botero MF, Healy NA, Hilsenbeck SG, Phillips GL, Chamness GC, Rimawi MF, Osborne CK, Schiff R. Different mechanisms for resistance to trastuzumab versus lapatinib in HER2-positive breast cancers--role of estrogen receptor and HER2 reactivation. Breast Cancer Res. 2011;13(6):R121. doi: 10.1186/bcr3067. Epub 2011 Nov 28. PMID 22123186
- [Background] Tan-Chiu E, Yothers G, Romond E, Geyer CE Jr, Ewer M, Keefe D, Shannon RP, Swain SM, Brown A, Fehrenbacher L, Vogel VG, Seay TE, Rastogi P, Mamounas EP, Wolmark N, Bryant J. Assessment of cardiac dysfunction in a randomized trial comparing doxorubicin and cyclophosphamide followed by paclitaxel, with or without trastuzumab as adjuvant therapy in node-positive, human epidermal growth factor receptor 2-overexpressing breast cancer: NSABP B-31. J Clin Oncol. 2005 Nov 1;23(31):7811-9. doi: 10.1200/JCO.2005.02.4091. PMID 16258083
- [Background] Slamon DJ, Leyland-Jones B, Shak S, Fuchs H, Paton V, Bajamonde A, Fleming T, Eiermann W, Wolter J, Pegram M, Baselga J, Norton L. Use of chemotherapy plus a monoclonal antibody against HER2 for metastatic breast cancer that overexpresses HER2. N Engl J Med. 2001 Mar 15;344(11):783-92. doi: 10.1056/NEJM200103153441101. PMID 11248153
- [Background] Rusnak DW, Lackey K, Affleck K, Wood ER, Alligood KJ, Rhodes N, Keith BR, Murray DM, Knight WB, Mullin RJ, Gilmer TM. The effects of the novel, reversible epidermal growth factor receptor/ErbB-2 tyrosine kinase inhibitor, GW2016, on the growth of human normal and tumor-derived cell lines in vitro and in vivo. Mol Cancer Ther. 2001 Dec;1(2):85-94. PMID 12467226